CLINICAL TRIAL: NCT02855489
Title: Condom Use Attitudes, Beliefs, and Behaviors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Boulder (Other)
Responsible Party: Principal Investigator, Angela Bryan, Professor, University of Colorado, Boulder
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: 13-0558
Record Dates: First submitted 2016-07-26; First posted 2016-08-04 (Estimated); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Condom Use
Keywords: Condom Use; HIV/STD; Intervention; Theory of Planned Behavior; Dismantling Study Design

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (7):
- Attitudes Only (Experimental): The attitudes condition targeted cognitive and affective attitudes by pairing attitudinal messages with pictures, and included an evaluative conditioning task.
  Interventions: Behavioral: Attitudes Only
- Norms Only (Experimental): The norms condition utilized a group-affirmation exercise, personalized feedback, and group norms in an attempt to greater condom use norms.
  Interventions: Behavioral: Norms Only
- Perceived Behavioral Control Only (Experimental): The PBC condition included a condom application video, lubrication instructions, condom negotiation videos, and a detailed description regarding purchasing condoms.
  Interventions: Behavioral: Perceived Behavioral Control Only
- Intentions Only (Experimental): The intentions condition utilized implementation intentions in order to create condom use intentions.
  Interventions: Behavioral: Intentions Only
- Three Constructs (Experimental): A three construct condition, which included attitudes, norms, and perceived behavioral control represented the core components of the TPB that are thought to work through intentions to result in behavior change.
  Interventions: Behavioral: Three Constructs
- Four Constructs (Experimental): A four construct condition (i.e., attitudes, norms, PBC, and intentions) was designed to represent the "full TPB model" intervention which we expected would be more successful than either the three-construct intervention or any of the single construct interventions.
  Interventions: Behavioral: Four Constructs
- No-Treatment, Control (No Intervention): A no-treatment control condition, which solely consisted of pretest and posttest assessments, was included. This allowed us to obtain important information about how the theoretical constructs in the TPB change over time (or do not) in the absence of an experimental manipulation.

INTERVENTIONS:
Behavioral: Attitudes Only
  Arms: Attitudes Only
Behavioral: Norms Only
  Arms: Norms Only
Behavioral: Perceived Behavioral Control Only
  Arms: Perceived Behavioral Control Only
Behavioral: Intentions Only
  Arms: Intentions Only
Behavioral: Three Constructs
  Arms: Three Constructs
Behavioral: Four Constructs
  Arms: Four Constructs

SUMMARY:
This study has three primary goals. First, to design distinct interventions that target the three core constructs of the Theory of Planned Behavior (i.e, attitudes, norms, and perceived behavioral control (PBC)). The second goal is to determine which combination of the Theory of Planned Behavior constructs is more successful at changing condom use behavior among college students. Finally, the investigators will examine the impact change in targeted constructs has on those not targeted by an intervention. The current study intends to empirically test how the constructs (i.e., attitudes, norms, PBC) in the Theory of Planned Behavior influence each other to increase condom use with college students.

DETAILED DESCRIPTION:
Theory allows researchers to systematically explain and predict health behavior by providing an organized framework to approach research questions; the importance of theory is particularly emphasized in meta-analyses demonstrating that interventions designed from the basis of health behavior theory are more successful than those that are not theory-based. The superiority of theory-based interventions has been established, but these meta-analyses do not answer the important questions of which theoretical constructs may be the "active ingredients" of change nor of how constructs in a particular theory may work separately versus in combination to produce the greatest amount of behavior change. Health interventions on the whole have only small to moderate effects on behavior change, and perhaps this is partly due to a lack of solid understanding of how key theoretical constructs influence each other to motivate behavior change. Often times when a theory is used as the basis for an intervention only a subset of the constructs seem to produce behavior change, which calls into question the sufficiency of our current theories for producing behavior change. One possible reason for this may be that current health behavior theories are really theories of behavioral prediction and not behavior change.

Health behavior theories are often used to inform intervention development-assuming that the same cognitive processes that successfully explain behavior are also the same processes that can be targeted to elicit behavior change. Past reviews show that theories like the Theory of Planned Behavior (TPB) explain 30%-50% of the variance in behavior, and when behavior change is the outcome the same predictors only produce small to moderate effects. However, it is unclear if the same predictors are working together in a similar way when using them to explain behavior versus creating behavior change. Currently, the same cognitive mechanisms are used to describe both processes, but those that explain behavior may not be the same ones that produce behavior change. There is very little literature that addresses how these processes may differ. A careful examination of the extent to which current theoretical constructs successfully produce behavior change individually or in combination may help clarify the optimal theoretical framework that should be utilized in behavior change interventions. Using the Theory of Planned Behavior (TPB) as the guiding theoretical framework, this study explores one way to experimentally determine how the constructs in the TPB influence each other and successfully produce health behavior change.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be 18 and older and must have had vaginal or anal intercourse at least once.

Exclusion Criteria:

* Prior research has indicated that the predictors of condom use are dramatically different in casual versus serious relationships and that condom use is extremely difficult to change among those in established long-term relationships. Thus, we will exclude participants if they indicate that they are in a relationship and they classify that relationship as someone they are "living with" or "married to".

Ages: 18 Years to 26 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 317 (Actual)
Dates: Start 2013-11; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Risky Sexual Behavior | Three Months
  Risky sexual behavior was a composite variable calculated using "how many times a participant had sex in the past 3 months" X "how many times they used a condom when having sex during those 3 months" (reverse coded). Higher scores indicated riskier sexual behavior.

SECONDARY OUTCOMES:
Condom Use | Three Months
  Condom use was measured by asking participants "In the past 3 months only, how much of the time have you used condoms when you've had sexual intercourse?" on a scale from 0% of the time to 100% of the time.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Reid AE, Aiken LS. Integration of five health behaviour models: common strengths and unique contributions to understanding condom use. Psychol Health. 2011 Nov;26(11):1499-520. doi: 10.1080/08870446.2011.572259. Epub 2011 Jun 28. PMID 21678166
- [Background] Glanz K, Bishop DB. The role of behavioral science theory in development and implementation of public health interventions. Annu Rev Public Health. 2010;31:399-418. doi: 10.1146/annurev.publhealth.012809.103604. PMID 20070207
- [Background] Glanz K, Maddock J. On judging models and theories: research and practice, psychology and public health. J Health Psychol. 2000 Mar;5(2):151-4. doi: 10.1177/135910530000500203. No abstract available. PMID 22049003
- [Background] Noar SM. Behavioral interventions to reduce HIV-related sexual risk behavior: review and synthesis of meta-analytic evidence. AIDS Behav. 2008 May;12(3):335-53. doi: 10.1007/s10461-007-9313-9. Epub 2007 Sep 21. PMID 17896176
- [Background] Godin G, Kok G. The theory of planned behavior: a review of its applications to health-related behaviors. Am J Health Promot. 1996 Nov-Dec;11(2):87-98. doi: 10.4278/0890-1171-11.2.87. PMID 10163601
- [Background] Webb TL, Sheeran P. Does changing behavioral intentions engender behavior change? A meta-analysis of the experimental evidence. Psychol Bull. 2006 Mar;132(2):249-68. doi: 10.1037/0033-2909.132.2.249. PMID 16536643
- [Derived] Montanaro EA, Kershaw TS, Bryan AD. Dismantling the theory of planned behavior: evaluating the relative effectiveness of attempts to uniquely change attitudes, norms, and perceived behavioral control. J Behav Med. 2018 Dec;41(6):757-770. doi: 10.1007/s10865-018-9923-x. Epub 2018 Apr 18. PMID 29671166